CLINICAL TRIAL: NCT06017375
Title: Patient Knowledge, Beliefs and Barriers to Hepatitis D Care; Single Site Observational Study
Brief Title: Patient Knowledge, Beliefs and Barriers to Hepatitis D Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 330645
Record Dates: First submitted 2023-08-17; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis, Delta
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire based intervention — Three validated questionnaires amended from hepatitis B to D (Chronic liver disease questionnaire, self-stigma scale and HBV virus knowledge scale) will be used.

SUMMARY:
A project to understand the determinants of health behaviour among those with chronic hepatitis D virus (HDV) infection, under the care of the viral hepatitis service at Kings College Hospital (KCH). This is to improve and implement pathways and patient information distribution to improve access to care in an ethnically diverse population living with HDV in the UK.

Kings college hospital NHS Foundation Trust is uniquely placed and serves a large diverse population from areas such as pan pacific Asia, Eastern Europe and regions in Africa, where English is not their first language. This diversity is also seen in other London Hospitals but less so in other parts of the UK.

DETAILED DESCRIPTION:
To understand the knowledge patients have around their diagnosis of hepatitis D which is considered a rare disease but the most aggressive form of viral hepatitis. In order to improve the management of hepatitis D, this research aims to identify the current knowledge patients have about their diagnosis, the information provided to them in their preferred language, how they feel about their diagnosis and the stigma attached. This research has been conducted in patients with other forms of viral hepatitis but not in patients living with hepatitis D. There is a lack of research in this area. With this research we aim to improve treatment pathways, access to care and to information.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years or older.
* HDV infection as diagnosed by high levels of anti-HDV immunoglobulin G (IgG) and immunoglobulin M (IgM), and confirmed by detection of HDV RNA in serum.
* Treated HDV infection
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Clinically significant medical or psychiatric illness in the past, present, or being evaluated, that may interfere with participant treatment, safety and assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with past or current hepatitis D virus infection
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
The overall patient understanding of Hepatitis D Virus diagnosis | 6 months
  Use of modified CLDQ - HBV survey. Scale of 1-7 with lower scores indicating worse outcomes
Describe overall patient knowledge around HDV | 6 months
  Modified HBV knowledge scale survey. Yes or No as options

SECONDARY OUTCOMES:
Describe stigma attached towards HDV | 6 months
  Use of modified Toronto HBV stigma questionnaire. Scale options are: never, rarely, sometimes, often, always
Understand satisfaction with communication regarding HDV care at KCH | 6 months
  Use of local viral hepatitis service questionnaire

IPD SHARING:
Plan to Share IPD: No